CLINICAL TRIAL: NCT00329719
Title: A Phase I/II Trial of Sorafenib and CCI-779 in Patients With Recurrent Glioblastoma
Brief Title: Sorafenib Tosylate and Temsirolimus in Treating Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00652; NCI-2009-00652 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000472240; NCCTG-N0572; N0572 (Other: Alliance for Clinical Trials in Oncology); N0572 (Other: CTEP); U10CA180821 (NIH); U10CA025224 (NIH)
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Sorafenib; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (sorafenib tosylate, temsirolimus) (Experimental): Patients receive sorafenib tosylate and temsirolimus as in Phase I.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Sorafenib Tosylate; Drug: Temsirolimus
- Group II (sorafenib tosylate, temsirolimus, surgery) (Experimental): Patients receive sorafenib tosylate PO BID on days 1-8 and temsirolimus IV over 30 minutes on day 1. Patients undergo surgery on day 8. After recovering from surgery, patients receive sorafenib tosylate and temsirolimus as in Phase I.
  Interventions: Procedure: Conventional Surgery; Other: Laboratory Biomarker Analysis; Drug: Sorafenib Tosylate; Drug: Temsirolimus
- Group III (sorafenib tosylate, temsirolimus, anti-VEGF) (Experimental): Patients who have received prior anti-VEGF therapy and are not undergoing surgery receive sorafenib tosylate and temsirolimus as in Phase I.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Sorafenib Tosylate; Drug: Temsirolimus

INTERVENTIONS:
Procedure: Conventional Surgery — Undergo surgery
  Arms: Group II (sorafenib tosylate, temsirolimus, surgery)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This phase I/II trial studies the side effects and best dose of temsirolimus when given together with sorafenib tosylate and to see how well they work in treating patients with glioblastoma that has come back. Sorafenib tosylate may stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as temsirolimus, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sorafenib tosylate and temsirolimus may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving sorafenib tosylate with temsirolimus may kill more tumor cells.

DETAILED DESCRIPTION:
Primary Objective -

Phase I (closed to accrual as of 01/11/2008):

To establish a maximum tolerable dose of temsirolimus in combination with sorafenib in patients with recurrent glioblastoma not receiving enzyme-inducing anticonvulsants (EIACs).

Phase II (closed to accrual as of 12/07/2012):

To assess the efficacy of temsirolimus and sorafenib in the treatment of recurrent glioblastoma in non-EIAC patients as measured by progression-free survival status at six months (PFS6).

Secondary Objectives -

Phase I (closed to accrual as of 01/11/2008):

I. To define the safety profile of temsirolimus and sorafenib in non-EIAC patients.

II. To assess the evidence of antitumor activity.

Phase II (closed to accrual as of 12/07/2012):

I. To assess the safety and toxicities of temsirolimus and sorafenib in the above-noted patient populations.

Outline: This is a multicenter, phase I, dose-escalation study followed by a phase II study.

Phase I (Arm A): Patients receive sorafenib orally (PO) twice daily (BID) on days 1-28 and temsirolimus intravenously (IV) over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of temsirolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Phase II: Patients are assigned to 1 of 3 treatment groups.

Group 1 (Arm B): Patients receive sorafenib and temsirolimus as in phase I at the MTD. (patients not undergoing surgery)

Group 2 (Arm C): Patients receive sorafenib PO BID on days 1-8 (15 doses) and temsirolimus IV at the MTD on day 1. Patients undergo surgery on day 8. (patients undergoing surgery) After recovering from surgery, patients receive sorafenib and temsirolimus as in phase I at the MTD.

Group 3 (Arm D): Patient receive sorafenib and temsirolimus as in phase I at the MTD. (patients who have received prior anti-vascular endothelial growth factor [VEGF] therapy and are not undergoing surgery)

Biopsy or resected tissue and blood are collected prior to treatment (usually at diagnosis) and analyzed for biomarkers. After completion of study treatment, patients are followed every 6 months for 5 years and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Central pathology review submission; this review is mandatory prior to registration to confirm eligibility; it should be initiated as soon after surgery as possible
* =< 2 prior systemic chemotherapy regimens
* Histological confirmation of a grade 4 astrocytoma (glioblastoma) or gliosarcoma, at primary diagnosis or recurrence by World Health Organization (WHO) criteria; central pathology review is mandatory prior to study entry to confirm eligibility
* Evidence of tumor progression by magnetic resonance imaging (MRI) or computed tomography (CT) scan following radiation therapy (RT) or following the most recent anti-tumor therapy
* Bidimensionally measurable or evaluable disease by MRI or CT scan
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* >= 12 weeks since the completion of RT
* Fixed or decreasing dose of corticosteroids (or no corticosteroids) >= 1 week prior to registration
* >= 1 week from minor surgery other than venous line placement and > 3 weeks from major surgery (except for patients undergoing tumor tissue acquisition)
* >= 4 weeks since prior cytotoxic chemotherapy (>= 6 weeks for nitrosoureas)
* >= 2 weeks from cytostatic chemotherapy such as tamoxifen, cis-retinoic acid, or thalidomide (address questions regarding such agents to study chair)
* White blood cells (WBC) >= 3,000/mm^3
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin (Hgb) >= 10 gm/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2.5 x ULN
* Creatinine =< 2.0 x ULN
* Serum cholesterol =< 350 mg/dL
* Serum triglycerides =< 400 mg/dL
* Willingness to provide the biologic specimens as required by the protocol; (please note that the willingness to participate pertains only to the patient and does not factor in the institution?s ability to participate in any part of the translational component)

Exclusion Criteria:

* Prior intratumoral chemotherapy (e.g., Gliadel or IL13-PE38QQR), stereotactic radiosurgery, or interstitial brachytherapy unless there is a separate lesion on MRI which is not part of the previous treatment field or there is proof of recurrent disease based on biopsy, MRI spectroscopy, or positron emission tomography (PET) scan
* Prior CCI-779, sorafenib, or other agents specifically targeting mammalian target of rapamycin (mTOR) or raf; patients receiving prior agents inhibiting VEGF or VEGF receptor (R) (prior anti-VEGF group) are eligible but: 1) must be at least four weeks from last treatment with the agent(s); and 2) must have recovered from any clinically relevant toxicities attributable to this agent(s)
* Evidence of bleeding diathesis or coagulopathy

  * Note: Patients on prophylactic anticoagulation therapy (e.g., low-dose warfarin) are eligible provided their coagulation parameter levels are as follows: prothrombin time (International Normalized Ratio [INR] of prothrombin time) < 1.1 x institutional upper limit of normal
  * Note: Patients on full-dose anticoagulants (e.g., warfarin) are eligible provided that both of the following criteria are met: a) the patient has an in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin, and b) the patient has no active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* International normalized ration (INR) > 1.5 (unless the patient is on full-dose warfarin)
* Receiving enzyme-inducing antiepileptic drugs (EIAEDs; e.g., phenytoin, fosphenytoin, carbamazepine, phenobarbital, or primidone) or any other potent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducer, such as rifampin or St. John?s wort
* Any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow pills
* Hypertension with systolic blood pressure of > 140 mmHg or diastolic pressure > 90 mmHg; however, patients with well-controlled hypertension are eligible
* Uncontrolled infection
* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Known hypersensitivity to any of the components of CCI-779 or sorafenib
* Other active malignancy
* Uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness/social situation that would preclude study compliance with study requirements
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive; HIV-positive patients on combination antiretroviral therapy are ineligible
* Receiving any investigational agents other than CCI-779 and sorafenib
* Significant intratumoral, intracerebral, or subarachnoid hemorrhage on baseline MRI or CT, or other history of significant intratumoral, intracerebral, or subarachnoid hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2006-03-24 (Actual); Primary Completion 2013-02-01 (Actual); Study Completion 2013-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Jaeckle, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (190):
- United States (190):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Saint Anthony Memorial Hospital, Effingham, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Minnesota Cooperative Group Outreach Program, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, Arm A: Phase I, Arm A, Dose Escalation
  Patients receive sorafenib orally (PO) twice daily (BID) on days 1-28 and temsirolimus intravenously (IV) over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of temsirolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  sorafenib tosylate: Given PO
  temsirolimus: Given IV
- Phase II, Arm B: Phase II, Arm B, Group I (patients not undergoing surgery)
  Patients receive sorafenib and temsirolimus at the MTD (25mg temsirolimus and 200mg sorafenib).
  sorafenib tosylate: Given PO
  temsirolimus: Given IV
- Phase II, Arm C: Phase II, Arm C, Group II (patients undergoing surgery)
  Patients receive sorafenib PO BID on days 1-8 (15 doses) and temsirolimus IV at the MTD on day 1. Patients undergo surgery on day 8. After recovering from surgery, patients receive sorafenib and temsirolimus as in phase I at the MTD (25mg temsirolimus and 200mg sorafenib).
  sorafenib tosylate: Given PO
  temsirolimus: Given IV
  conventional surgery: Undergo surgery
- Phase II, Arm D: Phase II, Arm D, Group III (patients who received prior anti-VEGF therapy)
  Patients receive sorafenib and temsirolimus as in phase I at the MTD (25mg temsirolimus and 200mg sorafenib).
  sorafenib tosylate: Given PO
  temsirolimus: Given IV
Period: Overall Study
Arm/Group | Phase I, Arm A | Phase II, Arm B | Phase II, Arm C | Phase II, Arm D
Started | 12 | 49 | 9 | 45
Completed | 12 | 49 | 9 | 44
Not Completed | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I, Arm A | Phase II, Arm B | Phase II, Arm C | Phase II, Arm D | Total
Number analyzed (Participants) | 12 | 49 | 9 | 45 | 115
Age, Continuous [Mean (Full Range); unit: years] | 53.8 [24 to 76] | 55.5 [24 to 74] | 58.4 [51 to 63] | 56.8 [29 to 75] | 56.0 [24 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 14 | 2 | 15 | 37
  Male | 6 | 35 | 7 | 30 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 0 | 3
  White | 12 | 46 | 7 | 45 | 110
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: The primary endpoint is the proportion of patients alive and progression-free 6 months after study treatment initiation.
  If more than 41 evaluable patients are accrued in group 1 or group 3, the additional patients will not be used to evaluate the decision rule for that group or otherwise used in any decision-making processes. However, they will be included in the final point and confidence interval estimates for that group.
  The 'success' probability, i.e., 6-month progression-free survival percentage, for each of group 1 and group 3 will be estimated as the number of evaluable patients still alive at 6 months divided by the total number of evaluable patients followed for at least 6 months. Ninety-five percent confidence intervals for the 'success' probability will be calculated according to the approach of Duffy and Santner.
  Progression is defined as a 25% increase in product of perpendicular diameters of contrast enhancement or mass or appearance of new lesions.
Time Frame: At 6 months
Measure: Number (95% Confidence Interval); unit: Proportion of Successes
Arm/Group | Phase I, Arm A | Phase II, Arm B | Phase II, Arm C | Phase II, Arm D
Number analyzed (Participants) | 0 | 41 | 0 | 41
Proportion of Successes |  | 17.1 [7.7 to 32.6] |  | 9.7 [3.2 to 24.1]

2. Secondary Outcome: Overall Survival
Description: The overall survival distribution will be estimated using the method of Kaplan-Meier.
Time Frame: From start of study registration to death due to any cause or until last follow-up, up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I, Arm A | Phase II, Arm B | Phase II, Arm C | Phase II, Arm D
Number analyzed (Participants) | 0 | 46 | 7 | 44
months |  | 6.55 [4.24 to 11.6] | 6.74 [2.63 to NA] — Value not reached | 3.93 [2.96 to 5.63]

3. Secondary Outcome: Objective Response, as Determined by a Neurological Exam, MRI, and/or CT Measurement
Description: The proportion of patients in each response category will be summarized and 90% confidence intervals calculated assuming that the incidence of response is binomially distributed.
Time Frame: Up to 5 years
Measure: Number (90% Confidence Interval); unit: proportion of patients
Arm/Group | Phase I, Arm A | Phase II, Arm B | Phase II, Arm C | Phase II, Arm D
Number analyzed (Participants) | 12 | 49 | 9 | 45
proportion of patients
  Progression | .5 [.25 to .75] | .24 [.15 to .37] | 0 [0 to 0] | .47 [.34 to .6]
  Stable | .5 [.25 to .75] | .59 [.46 to .71] | .89 [.57 to .99] | .42 [.3 to .56]
  Regression | 0 [0 to 0] | .06 [.02 to .15] | 0 [0 to 0] | .022 [.001 to .1]
  Partial Response | 0 [0 to 0] | 0.02 [.001 to .09] | 0 [0 to 0] | 0 [0 to 0]
  Complete Response | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Unknown/Not Evaluated | 0 [0 to 0] | .08 [.03 to .18] | .11 [.01 to .43] | .09 [.03 to .19]

4. Secondary Outcome: Progression-free Survival
Description: Kaplan-Meier survival curves will be used to estimate progression-time distributions.
Time Frame: Time from study registration to date of disease progression or last follow-up, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I, Arm A | Phase II, Arm B | Phase II, Arm C | Phase II, Arm D
Number analyzed (Participants) | 0 | 46 | 9 | 44
months |  | 2.71 [2.20 to 3.98] | 4.34 [2.63 to NA] — value not reached | 1.87 [1.48 to 2.23]

ADVERSE EVENTS:
Groups:
- Phase I, Arm A: Patients receive sorafenib orally (PO) twice daily (BID) on days 1-28 and temsirolimus intravenously (IV) over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of temsirolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  sorafenib tosylate: Given PO
  temsirolimus: Given IV
- Phase II, Arm B: Patients receive sorafenib and temsirolimus at the MTD (25mg temsirolimus and 200mg sorafenib).
  sorafenib tosylate: Given PO
  temsirolimus: Given IV
- Phase II, Arm C: Patients receive sorafenib PO BID on days 1-8 (15 doses) and temsirolimus IV at the MTD on day 1. Patients undergo surgery on day 8. After recovering from surgery, patients receive sorafenib and temsirolimus as in phase I at the MTD (25mg temsirolimus and 200mg sorafenib).
  sorafenib tosylate: Given PO
  temsirolimus: Given IV
  conventional surgery: Undergo surgery
- Phase II, Arm D: Patients receive sorafenib and temsirolimus as in phase I at the MTD (25mg temsirolimus and 200mg sorafenib).
  sorafenib tosylate: Given PO
  temsirolimus: Given IV
Arm/Group | Phase I, Arm A | Phase II, Arm B | Phase II, Arm C | Phase II, Arm D
Serious Adverse Events (participants affected / at risk) | 3/12 | 15/49 | 3/9 | 11/45
Other Adverse Events (participants affected / at risk) | 12/12 | 48/49 | 9/9 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Arm A (N=12) | Phase II, Arm B (N=49) | Phase II, Arm C (N=9) | Phase II, Arm D (N=45)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bone infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infective myositis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Opportunistic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 4 (4) | 0 (0) | 3 (3)
Serum cholesterol increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Arm A (N=12) | Phase II, Arm B (N=49) | Phase II, Arm C (N=9) | Phase II, Arm D (N=45)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 9 (14) | 28 (82) | 5 (18) | 22 (36)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 4 (4) | 1 (4) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (9) | 11 (17) | 4 (7) | 8 (10)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 11 (20) | 1 (2) | 10 (15)
Diarrhea (Gastrointestinal disorders) | 5 (11) | 21 (46) | 5 (39) | 15 (23)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 10 (14) | 0 (0) | 11 (14)
Nausea (Gastrointestinal disorders) | 2 (7) | 20 (30) | 1 (28) | 14 (19)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 10 (12) | 1 (3) | 7 (7)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (3)
Fatigue (General disorders) | 11 (24) | 46 (135) | 9 (49) | 39 (72)
Fever (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gait abnormal (General disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abdominal infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Bone infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 12 (26) | 2 (4) | 10 (15)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (3) | 0 (0) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 2 (7) | 12 (23) | 2 (2) | 9 (15)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 2 (3)
CD4 lymphocytes decreased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (7) | 0 (0) | 3 (6)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 3 (6) | 7 (9) | 2 (6) | 5 (5)
Lymphocyte count decreased (Investigations) | 0 (0) | 4 (6) | 0 (0) | 8 (13)
Neutrophil count decreased (Investigations) | 4 (6) | 11 (21) | 4 (14) | 5 (7)
Platelet count decreased (Investigations) | 7 (12) | 36 (70) | 7 (49) | 36 (65)
Serum cholesterol increased (Investigations) | 7 (13) | 23 (55) | 5 (15) | 25 (40)
Weight loss (Investigations) | 1 (1) | 2 (2) | 2 (6) | 8 (10)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 21 (42) | 5 (28) | 27 (38)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 16 (25) | 2 (3) | 14 (25)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 10 (11) | 1 (1) | 6 (9)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 1 (2) | 6 (7)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 2 (2) | 7 (14)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (3) | 13 (24) | 2 (2) | 15 (29)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2) | 5 (9) | 1 (1) | 5 (6)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 5 (8) | 0 (0) | 6 (8)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Serum triglycerides increased (Metabolism and nutrition disorders) | 8 (12) | 21 (51) | 4 (13) | 23 (40)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (11) | 0 (0) | 3 (3)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 1 (2) | 0 (0)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 5 (5) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (4) | 12 (27) | 6 (32) | 14 (18)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 7 (15) | 2 (5) | 5 (7)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 5 (9)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 5 (18) | 1 (2) | 3 (4)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (5)
Depression (Psychiatric disorders) | 0 (0) | 5 (5) | 1 (2) | 1 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 8 (17) | 0 (0) | 2 (3)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (2) | 4 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (4) | 5 (10) | 1 (1) | 2 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 3 (4) | 6 (13) | 0 (0) | 6 (10)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (12) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 4 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (6) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 8 (11) | 27 (65) | 7 (11) | 20 (34)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (3) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 23 (39) | 4 (7) | 19 (32)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less